CLINICAL TRIAL: NCT06841029
Title: Management of Nausea and Vomiting in Pregnancy and Hyperemesis Gravidarum: Evaluation of Clinical Practices in Five Maternity Hospitals in Île-de-France
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0051_MATERNITE_
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: He Study Focuses on Evaluating Current Clinical Practices Rather Than Testing an Intervention
Keywords: NVP, hyperemesis gravidarum, clinical practices, adequacy, recommendations,CNGOF
MeSH Terms: conditions — Hyperemesis Gravidarum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Midwives: Midwives involved in the care of patients suffering from nausea and vomiting of pregnancy and hypermesis gravidarum
- Obstetrician-Gynecologists: Obstetrician-Gynecologists involved in the care of patients suffering from nausea and vomiting of pregnancy and hypermesis gravidarum
- Gynecology-Obstetrics Interns: Gynecology-Obstetrics involved in the care of patients suffering from nausea and vomiting of pregnancy and hypermesis gravidarum

SUMMARY:
This clinical trial aims to evaluate the adequacy of healthcare professionals' clinical practices regarding nausea and vomiting in pregnancy (NVP) and hyperemesis gravidarum (HG) with the recommendations of the National College of French Obstetricians and Gynecologists (CNGOF). The study involves 117 participants and follows an observational, cross-sectional, multicenter study design conducted in five maternity hospitals in Île-de-France.

ELIGIBILITY:
Inclusion Criteria:

* Midwives, obstetrician-gynecologists, and gynecology-obstetrics interns working in the labor and delivery units, high-risk pregnancy units, and obstetric-gynecological emergency units of the five selected maternity hospitals.

Exclusion Criteria:

* Midwives or doctors in training (student midwives or medical externs)
* Midwives and obstetrician-gynecologists working in private practice

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted of 117 healthcare professionals from five maternity hospitals in Île-de-France, of which 104 responses were usable. The participants included:
  68 midwives (65.4%)
  27 obstetrician-gynecologists (26%)
  9 gynecology-obstetrics interns (8.6%)
  The distribution across hospitals was as follows:
  Center A: 45 respondents (21 midwives, 17 obstetrician-gynecologists, 7 interns)
  Center B: 17 respondents (all midwives)
  Center C: 15 respondents (12 midwives, 3 obstetrician-gynecologists)
  Center D: 15 respondents (9 midwives, 4 obstetrician-gynecologists, 2 interns)
  Center E: 12 respondents (9 midwives, 3 obstetrician-gynecologists)
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage of healthcare professionals whose management of NVP and HG aligns with CNGOF recommendations. | data collection period: October 2023-March 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Saint-Denis, Saint-Denis, France

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36150647/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26358678/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25830549/